CLINICAL TRIAL: NCT07055607
Title: A Two-year Prospective, Observational Study of Wegovy in Real-world Clinical Practice
Acronym: PILLAR
Status: Recruiting | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-8189; U1111-1308-1428 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-06-13; First posted 2025-07-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — semaglutide

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Wegovy®: Participants will be treated with Wegovy according to the local labels in Spain, Switzerland and the United Kingdom (UK).
  Interventions: Drug: Semaglutide

INTERVENTIONS:
Drug: Semaglutide — Participants will be treated with commercially available Wegovy according to routine clinical practice and is purely at the discretion of the treating physician. Only individuals receiving Wegovy reimbursed by the healthcare system in their respective countries are included in the study.
  Other Names: Wegovy®

SUMMARY:
This observational study will explore how Wegovy® (Semaglutide) is used in everyday situations, how it might affect things like weight, body mass index (BMI) and waist circumference, and what kind of impact it could have on overall quality of life. The overall purpose of this study is to understand how Wegovy impacts weight when used as part of regular medical care. Participants will be treated with Wegovy as prescribed to the participant by their doctor, in accordance with normal clinical practice. The study will last for about two years.

ELIGIBILITY:
Inclusion criteria:

* Signed consent obtained before any study-related activities (study-related activities are any pro-cedure related to recording of data according to the protocol).
* Are eligible for Wegovy and are due to initiate treatment for the first time within the study period; the decision to initiate treatment with commercially available Wegovy has been made by the patient/Legally Acceptable Representative (LAR) and the treating physician before and independently from the decision to include the patient in this study.
* Male or female, age above or equal to 18 years at time of signing informed consent.
* Have at least one reported weight measurement documented at baseline or within 28 days prior to baseline.
* Participants must be able to complete the electronic patient reported outcome (ePRO) questionnaires on a compatible electronic device with internet access.
* Fulfil the respective reimbursement criteria in the visit prior to / at baseline in Switzerland and United Kingdom (UK).

Exclusion criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study.
* Presence of a documented refusal or unwillingness to participate in research.
* Previous treatment with other obesity management pharmacotherapy or any glucagon like pep-tide-1 (GLP- 1) receptor agonist up to 90 days prior to baseline in Switzerland and UK.
* Previous treatment with other obesity management pharmacotherapy or any GLP- 1 receptor agonist up to 30 days prior to baseline in Spain.
* Pregnant or women of childbearing potential and not using a highly effective contraceptive method.
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation with the study requirements.
* Individuals who have reported plans to move out in the next 12 months to an area not serviced by their current site.
* Personal or family history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia syndrome type 2 (MEN 2) in Spain and UK.
* Participant has had a prior serious allergic reaction to semaglutide or any of the ingredients in Wegovy.
* Have had Saxenda reimbursed by basic mandatory health insurance for a cumulative period of more than 12 months prior to baseline in Switzerland.
* Documented history of diabetes mellitus type 1 and type 2 in Spain.
* Presence of diabetic complications and/or at risk of hypoglycaemia (with a documented history of frequent hypoglycaemia) in Spain.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be treated with Wegovy according to the local labels in Spain, Switzerland and the United Kingdom (UK).
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Estimated)
Dates: Start 2025-11-21 (Actual); Primary Completion 2027-10-25 (Estimated); Study Completion 2027-10-25 (Estimated)

PRIMARY OUTCOMES:
Absolute change in body weight (kilograms [kg]) | From baseline (0 months) to the end of observation (24 months)
  Measured in kg.
Percentage change in body weight (percentage [%]) | From baseline (0 months) to the end of observation (24 months)
  Measured in %.

SECONDARY OUTCOMES:
Absolute change in waist circumference (centimeters [cm]) | From baseline (0 months) to the end of observation (24 months)
  Measured in cm.
Absolute change in waist-to-height ratio | From baseline (0 months) to the end of observation (24 months)
  Measured as ratio.
Percentage change in waist circumference (%) | From baseline (0 months) to the end of observation (24 months)
  Measured in %.
Number of participants who achieve greater than or equal to (>=) 5 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Measured as count of participants.
For Switzerland: Number of participants who achieve >=7 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (22 months)
  Measured as count of participants.
Number of participants who achieve >=10 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Measured as count of participants.
For Switzerland: Number of participants who achieve >=12 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (22 months)
  Measured as count of participants.
Number of participants who achieve >=15 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Measured as count of participants.
Number of participants who achieve >=20 percent body weight reduction (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Measured as count of participants.
Change in percentage of participant in each Body Mass Index (BMI) category | From baseline (0 months) to the end of observation (24 months)
  Measured as count of participants.
Change in High Density Lipoprotein (HDL) Cholesterol (milligrams per decilitre [mg/dL]) | From baseline (0 months) to the end of observation (24 months)
  Measured in mg/dL.
Change in HDL Cholesterol (millimoles per litre [mmol/L]) | From baseline (0 months) to the end of observation (24 months)
  Measured in mmol/L.
Change in Low Density Lipoprotein (LDL) Cholesterol (mg/dL) | From baseline (0 months) to the end of observation (24 months)
  Measured in mg/dL.
Change in LDL Cholesterol (mmol/L) | From baseline (0 months) to the end of observation (24 months)
  Measured in mmol/L.
Change in Very Low Density Lipoprotein (VLDL) Cholesterol (mg/dL) | From baseline (0 months) to the end of observation (24 months)
  Measured in mg/dL.
Change in VLDL Cholesterol (mmol/L) | From baseline (0 months) to the end of observation (24 months)
  Measured in mmol/L.
Change in Free Fatty Acid (FFA) (mmol/L) | From baseline (0 months) to the end of observation (24 months)
  Measured in mmol/L.
Change in Triglycerides (mg/dL) | From baseline (0 months) to the end of observation (24 months)
  Measured in mg/dL.
Change in Triglycerides (mmol/L) | From baseline (0 months) to the end of observation (24 months)
  Measured in mmol/L.
Change in Glycated Haemoglobin (HbA1c) (%) | From baseline (0 months) to the end of observation (24 months)
  Measured in %.
Change in systolic blood pressure | From baseline (0 months) to the end of observation (24 months)
  Measured in millimeter of mercury (mmHg).
Change in diastolic blood pressure | From baseline (0 months) to the end of observation (24 months)
  Measured in mmHg.
Percentage change in the prevalence of obesity-related conditions | From baseline (0 months) to the end of observation (24 months)
  Obesity-related conditions will be assessed as Yes/No in the following categories: Myocardial infarction (MI), Stroke, Heart failure with reduced Ejection Fraction (HFrEF) and Heart Failure with preserved Ejection Fraction (HFpEF), Atherosclerotic cardiovascular disease (ASCVD) defined as at least one of coronary artery disease, peripheral artery disease, cerebrovascular disease and atherosclerosis, Metabolic dysfunction-associated steatotic liver disease (MASLD), Metabolic dysfunction-associated steatohepatitis (MASH), Chronic kidney disease (CKD), Obstructive sleep apnoea, Poly-cystic ovary syndrome (PCOS), Infertility, Urinary incontinence, Lower back pain, Knee / hip oste-oarthritis, Musculoskeletal pain, Asthma, Chronic Obstructive Pulmonary Disease (COPD), Clini-cian-diagnosed mood disorder, Clinician-diagnosed eating disorder.
Percentage change in the total daily dosage of concomitant drugs (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Total daily dosage of concomitant drugs were assessed as Yes/No among the following: Antidiabetic medication, Antihypertensive medication, Lipid-lowering medication, Pain medica-tion, Psychotropic medication, Antithrombotic agents, Thyroid hormone medication, Proton pump inhibitor.
Percentage change in the usage of additional treatments for weight loss (Yes/No) | From baseline (0 months) to the end of observation (24 months)
  Usage of additional treatments for weight loss will be assessed as Yes/No among the following: Bariatric surgery, Clinical practice / healthcare-provided diet plan, Alternative diet plan, Exercise regime, Behavioural and alternative therapy, Digital health app.
Median time to Wegovy® maintenance dose | From baseline to the date of reported maintenance dose during the observation period (24 months)
  Measured in weeks.
Median time to each Wegovy® dose escalation | Date from the start of the previous dose to the date of each subsequent escalation during the observation period (24 months)
  Measured in weeks.
Maximum dose of Wegovy® for weight management | After baseline to any given time during the observation period (24 months)
  Measured in milligrams (mg).
For UK and Spain: Change in percentage of participants on Wegovy® with each of drug-related adverse reaction | From baseline (0 months) to the end of observation (24 months)
  Measured as percentage of participants.
Median persistence time of Wegovy® treatment | From baseline (0 months) to the end of observation (24 months)
  Measured in weeks.
Change in percentage of participants who discontinued | From baseline (0 months) to the end of observation (24 months)
  Measured as percentage of participants.
Percentage of participants who discontinued/withdrawn | From baseline (0 months) to the end of observation (24 months)
  Measured as percentage of participants. Reason for discountinued/withdrawn due to Lack of efficacy as per reimbursement criteria (UK, CH only), Lack of efficacy as per clinical judgment, Lack of efficacy as per subject's judgment, Non-serious gastro intestinal event (nausea, vomiting, diarrhea, constipation and/or abdominal pain), Adverse reaction ((AR) not otherwise specified in the listed reasons), Patient's request, Pregnancy,Financial constraints (cost of medication, change in eligibility for reimbursement) (CH and ES only), Reaching a BMI of less than (<) 25 kilograms per meter square (kg/m^2), death and other.
For Switzerland: Percentage of participants who continued under reimbursement by basic mandatory health insurance (Yes/No) | From baseline (0 months) to the end of observation (22 months)
  Measured as percentage of participants.
For Switzerland: Percentage of participants who switched to out-of-pocket payment (or any other arrangement) (Yes/No) | From baseline (0 months) to the end of observation (22 months)
  Measured as percentage of participants.
For Switzerland: Percentage of participants who stopped treatment (Yes/No) | From baseline (0 months) to the end of observation (22 months)
  Measured as percentage of participants.
For Spain: Percentage of participants who have continued under out-of-pocket payment (Yes/No) | From baseline (0 months) to the end of observation (12 months)
  Measured as percentage of participants.
For Spain: Percentage of participants who have switched to reimbursement by the Public Health System (Yes/No) | From baseline (0 months) to the end of observation (12 months)
  Measured as percentage of participants.
For Switzerland: Change in percentage of participants fulfilling the necessary weight loss reimbursement criteria | From baseline (0 months) to the end of observation (22 months)
  Measured as percentage of participants.
Absolute change in the EuroQoL-5-Dimension (5-Level) (EQ-5D-5L) | From baseline (0 months) to the end of observation (24 months)
  EQ-5D-5L consists of 2 components, EQ-5D descriptive system and EQ visual analogue scale (EQ-VAS). EQ-5D 5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension will have 5 levels: no, slight, moderate, severe and extreme problems. Respondent is asked to indicate the health state by ticking the box next to the most appropriate statement in each of the five dimensions. Decision will result in a 1-digit number that expresses the level for that dimension. Digits for five dimensions can be combined into a 5-digit number that describes patient's health state. EQ-5D health states can be converted into a single summary number (index value) which will reflect how good/bad a health state is according to valuation set in general population of a country/region. Index score records an average health status according to dimensions using an algorithm,ranges 0-1 with higher score indicating better health status.
Absolute change in the EQ Visual Analogue Score (EQ-VAS) | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. The EQ-VAS will record the respondent's self-rated health on a vertical visual analogue scale. The scale is numbered from 0 to 100, with lower score indicating worst health and higher score indicating best health.
Absolute change in the Adelphi Adherence Questionnaire (ADAQ) score | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. ADAQ is an 11-item instrument that measures adherence to medication. The instrument includes 4 items that assess adherence behaviours and 7 items that assess drivers of non adherence. Each item yields a score ranging from 0 to 4 and item scores are then averaged to produce the ADAQ score. The ADAQ score is a measure of medication adherence ranging from 0 to 4, with lower scores representing greater adherence.
Absolute change in treatment satisfaction questionnaire for medication 9 (TSQM-9) domain scores | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. TSQM-9 is a 9-item instrument that measures a patient's satisfaction with their medication. The instrument assesses three domains: effectiveness, convenience and global satisfaction. Each domain will produce a score ranging from 0 to 100, with higher scores reflecting higher satisfaction on that domain.
Absolute change in percentage of work time missed (absenteeism) due to weight problem using Work Productivity and Activity Impairment Questionnaire (WPAI) | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. WPAI is a self-administered instrument used to assess the impact of disease on work productivity and regular activities during the past seven days. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Absolute change in percentage of time impaired while working (presenteeism) due to weight problem using WPAI | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. WPAI is a self-administered instrument used to assess the impact of disease on work productivity and regular activities during the past seven days. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.
Absolute change in percentage of activity impairment due to weight problem using WPAI | From baseline (0 months) to the end of observation (24 months)
  Measured as score points. WPAI is a self-administered instrument used to assess the impact of disease on work productivity and regular activities during the past seven days. WPAI outcomes are expressed as impairment percentages (0-100), with higher numbers indicating greater impairment and less productivity, that is, worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (8):
- Switzerland (2):
  - Hôpitaux Universitaires de Genève (HUG), Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
- United Kingdom (6):
  - Sandwell Health Campus, West Bromwich, West Midlands
  - Barnsley Hospital, Barnsley
  - Hull Royal Infirmary, Hull
  - Evelina London Children's Hospital, London
  - Luton and Dunstable University Hospital, Luton
  - St George's Hospital, Tooting

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com